CLINICAL TRIAL: NCT02787005
Title: Phase II Trial of Pembrolizumab (MK-3475) in Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC) (KEYNOTE-199)
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC)(MK-3475-199/KEYNOTE-199)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-199; 163366 (Registry Identifier: JAPIC-CTI); MK-3475-199 (Other: MSD); KEYNOTE-199 (Other: MSD); 2015-003644-40 (EudraCT Number)
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: PD-L1 positive with measurable disease (Experimental): Participants with programmed cell death ligand 1 (PD-L1)-positive, measurable disease receive pembrolizumab 200 mg via intravenous infusion on Day 1 of every 3-week cycle for up to 2 years.
  Interventions: Biological: Pembrolizumab
- Cohort 2: PD-L1 negative with measurable disease (Experimental): Participants with PD-L1 negative, measurable disease receive pembrolizumab 200 mg via intravenous infusion on Day 1 of every 3-week cycle for up to 2 years.
  Interventions: Biological: Pembrolizumab
- Cohort 3: Bone metastases with non-measurable disease (Experimental): Participants with bone metastases and non-measurable disease receive pembrolizumab 200 mg via intravenous infusion on Day 1 of every 3-week cycle for up to 2 years.
  Interventions: Biological: Pembrolizumab
- Cohort 4: RECIST 1.1-measureable disease (Experimental): Participants with Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)-measureable disease receive pembrolizumab 200 mg via intravenous infusion on Day 1 of every 3-week cycle for up to 2 years.
  Interventions: Biological: Pembrolizumab
- Cohort 5: Bone metastases only or bone-predominant disease (Experimental): Participants with bone metastases only or bone-predominant disease receive pembrolizumab 200 mg via intravenous infusion on Day 1 of every 3-week cycle for up to 2 years.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This is a study of pembrolizumab (MK-3475) in participants with metastatic castration-resistant prostate cancer (mCRPC). Participants will be enrolled into one of five cohorts: Cohort 1 (participants with programmed cell death ligand 1 [PD-L1]-positive, measurable disease), Cohort 2 (participants with PD-L1 negative, measurable disease), Cohort 3 (participants with bone-metastases and non-measurable disease) post-chemotherapy, Cohort 4 (participants with Response Evaluation Criteria in Solid Tumors version 1.1- [RECIST 1.1]-measureable disease) and Cohort 5 (participants with bone metastases only or bone-predominant disease) pre-chemotherapy.

DETAILED DESCRIPTION:
Participants with mCRPC previously treated with docetaxel-based chemotherapy in Cohorts 1 to 3 will receive monotherapy with pembrolizumab. Chemotherapy-naïve subjects with mCRPC either having failed or showing signs of failure with enzalutamide in Cohorts 4 and 5 will receive pembrolizumab monotherapy in addition to their current regimen of enzalutamide. In all cohorts, pembrolizumab administration will occur on Day 1 of each 3-week dosing cycle and will continue for a maximum of 35 cycles (approximately 2 years) unless specific withdrawal/discontinuation criteria are met. Participants who discontinue after 35 infusions of pembrolizumab for reasons other than disease progression or intolerability, or who discontinue after attaining a complete response may be eligible for up to 17 additional infusions (approximately 1 year) after they have experienced disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology. Disease must be either metastatic or locally confined inoperable disease that cannot be treated with definitive intent (no chance for a curative intervention).
* Has supplied tumor tissue from a newly obtained biopsy or a biopsy obtained ≤12 months prior to study start and an archival specimen, if available, from a site not previously irradiated. Participants in Cohorts 1, 2, and 4 with visceral/measurable lesions must provide a newly obtained biopsy performed after the last line of systemic therapy or a biopsy obtained ≤12 months prior to study start and an archival specimen, if available. Participants in Cohorts 3 and 5 must at least provide an archival specimen.

For Cohorts 1, 2, and 3 only:

* Has been treated with:
* At least 1 targeted endocrine therapy (defined as second generation antiandrogen therapies that include but are not limited to abiraterone acetate with prednisone, enzalutamide, and next generation targeted agents such as ARN-509).
* At least 1 regimen/line of chemotherapy that contained docetaxel.
* No more than 2 chemotherapy regimens.
* No more than 3 regimens/lines of the aforementioned treatments (having failed/progressed on chemotherapy and targeted endocrine therapy).

For Cohorts 4 and 5 only:

* Failing or showing early signs of failure on current pre-chemotherapy enzalutamide treatment as defined by Prostate Cancer Working Group 3 (PCWG3) guidelines. Participants can have failed prior abiraterone treatment before current enzalutamide treatment. Participants must have had a clinically meaningful response to enzalutamide treatment. Enzalutamide must have been initiated no less than 4 weeks prior to the first dose of trial treatment and be continued throughout the study.

For All Cohorts:

* Has documented prostate cancer progression within 6 months prior to screening, as determined by the Investigator, by means of one of the following: 1) PSA progression as defined by a minimum of 3 rising PSA levels with an interval of ≥1 week between each assessment where the PSA value at screening should be ≥2 ng/mL, OR, 2) Radiographic disease progression in soft tissue or bone with or without PSA progression
* Has ongoing androgen deprivation with total serum testosterone <50 ng/dL (<2.0 nM).
* Participants receiving bone resorptive therapy (including but not limited to bisphosphonate or Receptor activator of nuclear factor kappa-B ligand [RANK-L inhibitor]) must have been on stable doses for ≥4 weeks prior to first dose of study drug.
* Has a performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Participants of reproductive potential must agree to use an adequate method of contraception, starting with the first dose of study drug through at least the time needed to eliminate each study intervention after the last dose of study intervention. The length of time required to continue contraception after the last dose of enzalutamide is 30 days.
* Demonstrates adequate organ function.

Exclusion Criteria:

For All Cohorts:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of study drug.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of study drug or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from AEs due to mAbs administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or external beam radiation therapy within 4 weeks prior to the first dose of study drug or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from AEs due to a previously administered agent.
* Has a known additional malignancy that has had progression or has required active treatment in the last 3 years. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has evidence of interstitial lung disease and/or a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has previously participated in any other pembrolizumab (MK-3475) trial, or received prior therapy with an anti-programmed cell death 1 (anti-PD-1, anti-PD ligand 1 [anti-PD-L1], and anti-PD-L2 [including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways]).
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Has received a live vaccine within 30 days of planned start of study drug. Any licensed coronavirus disease 2019 (COVID-19) vaccine (including for Emergency use) in a particular country is allowed in the study as long as they are messenger ribonucleic acid (mRNA) vaccines, adenoviral vaccines, or inactivated vaccines. Investigational vaccines (ie, those not licensed or approved for Emergency Use) are not allowed.

For Cohorts 4 and 5 only:

* Has received prior chemotherapy (e.g., docetaxel) for mCPRC.
* Has any condition (cardiac, neurologic, absorption) other than clinically failing or showing early signs of failure on enzalutamide treatment that would require imminent discontinuation of enzalutamide treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Antonarakis ES, Piulats JM, Gross-Goupil M, Goh J, Ojamaa K, Hoimes CJ, Vaishampayan U, Berger R, Sezer A, Alanko T, de Wit R, Li C, Omlin A, Procopio G, Fukasawa S, Tabata KI, Park SH, Feyerabend S, Drake CG, Wu H, Qiu P, Kim J, Poehlein C, de Bono JS. Pembrolizumab for Treatment-Refractory Metastatic Castration-Resistant Prostate Cancer: Multicohort, Open-Label Phase II KEYNOTE-199 Study. J Clin Oncol. 2020 Feb 10;38(5):395-405. doi: 10.1200/JCO.19.01638. Epub 2019 Nov 27. PMID 31774688
- [Result] Graff JN, Hoimes CJ, Gerritsen WR, Vaishampayan UN, Elliott T, Hwang C, Ten Tije AJ, Omlin A, McDermott RS, Fradet Y, Tagawa ST, Kilari D, Ferrario C, Uemura H, Jones RJ, Fukasawa S, Peer A, Niu C, Poehlein CH, Qiu P, Suttner L, de Wit R, Schloss C, de Bono JS, Antonarakis ES. Pembrolizumab plus enzalutamide for metastatic castration-resistant prostate cancer progressing on enzalutamide: cohorts 4 and 5 of the phase 2 KEYNOTE-199 study. Prostate Cancer Prostatic Dis. 2025 Jun;28(2):411-418. doi: 10.1038/s41391-024-00865-5. Epub 2024 Aug 12. PMID 39134652
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Male participants at least 18 years of age with Metastatic Castration-resistant Prostate Cancer (mCRPC) were screened for enrollment in the study. Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Cohort 1: PD-L1 Positive With Measurable Disease: Participants with Programmed Cell Death 1 Receptor (PD-L1)-positive, measurable disease received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of every 3-week cycle for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Cohort 2: PD-L1 Negative With Measurable Disease: Participants with PD-L1 negative, measurable disease received pembrolizumab 200 mg via IV infusion on Day 1 of every 3-week cycle for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Cohort 3: Bone Metastases With Non-measurable Disease: Participants with bone metastases and non-measurable disease received pembrolizumab 200 mg via IV infusion on Day 1 of every 3-week cycle for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Cohort 4: RECIST 1.1-measureable Disease: Participants with RECIST 1.1-measureable disease received pembrolizumab 200 mg via IV infusion on Day 1 of every 3-week cycle for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab with SD or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Cohort 5: Bone Metastases Only or Bone-predominant Disease: Participants with bone metastases only or bone-predominant disease received pembrolizumab 200 mg via IV infusion on Day 1 of every 3-week cycle for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab with SD or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Period: Overall Study
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease
Started | 133 | 69 | 58 | 81 | 47
Treated | 133 | 67 | 58 | 81 | 45
Received 2nd Course | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 133 | 69 | 58 | 81 | 47
Not completed — Adverse Event | 24 | 9 | 9 | 7 | 2
Not completed — Death | 100 | 53 | 48 | 69 | 38
Not completed — Sponsor Decision | 7 | 4 | 0 | 4 | 5
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 1
Not completed — Screen Failure | 0 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: PD-L1 Positive With Measurable Disease: Participants with PD-L1-positive, measurable disease received pembrolizumab 200 mg via IV infusion on Day 1 of every 3-week cycle for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab with SD or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Total
Number analyzed (Participants) | 133 | 69 | 58 | 81 | 47 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (7.6) | 68.6 (7.2) | 69.4 (7.1) | 73.1 (8.4) | 69.7 (9.5) | 69.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 133 | 69 | 58 | 81 | 47 | 388
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 1 | 3 | 3 | 14
  Not Hispanic or Latino | 121 | 55 | 55 | 76 | 44 | 351
  Unknown or Not Reported | 9 | 10 | 2 | 2 | 0 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 6 | 7 | 5 | 2 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 3 | 3 | 11
  White | 109 | 52 | 48 | 70 | 42 | 321
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 8 | 10 | 2 | 2 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Cohort 1, Cohort 2, Cohort 4 and Cohorts 1 and 2 Combined)
Description: ORR was defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 by central imaging vendor. Per protocol, analysis for this outcome measure was conducted in Cohorts 1 and 2 combined, as well as in Cohorts 1, 2, and 4 separately for the first course of treatment.
Time Frame: Up to ~52 months
Population: Analysis population was the All Subjects as Treated (ASaT) which consisted of all allocated participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort 1: PD-L1 Positive With Measurable Disease: Participants with PD-L1-positive, measurable disease received pembrolizumab 200 mg via IV infusion
- Cohort 2: PD-L1 Negative With Measurable Disease: Participants with PD-L1 negative, measurable disease received pembrolizumab 200 mg via IV infusion
- Cohort 4: RECIST 1.1-measureable Disease: Participants with RECIST 1.1-measureable disease received pembrolizumab 200 mg via IV infusion
- Cohorts 1 and 2 Combined: Participants with PD-L1-positive, measurable disease or PD-L1 negative, measurable disease received pembrolizumab 200 mg via IV infusion
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohorts 1 and 2 Combined
Number analyzed (Participants) | 133 | 67 | 81 | 200
Percentage of Participants | 6.0 [2.6 to 11.5] | 3.0 [0.4 to 10.4] | 12.3 [6.1 to 21.5] | 5.0 [2.4 to 9.0]

2. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The percentage of participants that experienced at least one AE for the first course of treatment was reported.
Time Frame: Up to ~52 months
Population: Analysis population was the ASaT which consisted of all allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of Participants
Groups:
- Cohort 3: Bone Metastases With Non-measurable Disease: Participants with bone metastases and non-measurable disease received pembrolizumab 200 mg via IV infusion
- Cohort 5: Bone Metastases Only or Bone-predominant Disease: Participants with bone metastases only or bone-predominant disease received pembrolizumab 200 mg via IV infusion
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease
Number analyzed (Participants) | 133 | 67 | 58 | 81 | 45
Percentage of Participants | 99.2 | 97.0 | 100.0 | 98.8 | 97.8

3. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The percentage of participants who discontinued study treatment during the first course of treatment due to an AE was reported.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease
Number analyzed (Participants) | 133 | 67 | 58 | 81 | 45
Percentage of Participants | 10.5 | 3.0 | 12.1 | 18.5 | 20.0

4. Secondary Outcome: Disease Control Rate (DCR) (By Each Cohort, Cohorts 1 and 2 Combined, Cohorts 1, 2, and 3 Combined, Cohorts 4 and 5 Combined)
Description: Percentage of participants who had CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions)or stable disease (SD; Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) for at least 6 months, by central imaging vendor where progressive disease (PD) in bone-only tumors were determined by radionuclide bone scan using Prostate Cancer Working Group (PCWG3) criteria and PD for all other tumors was determined using RECIST 1.1. Per protocol, analysis for this outcome measure was conducted in Cohorts 1 and 2 combined, Cohorts 1,2, and 3 combined, Cohorts 4 and 5 combined well as in Cohorts 1 to 5 separately for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohorts 1, 2, and 3 Combined: Participants with PD-L1-positive, measurable disease, PD-L1 negative, measurable disease or bone metastases and non-measurable disease received pembrolizumab 200 mg via IV infusion
- Cohorts 4 and 5 Combined: Participants with RECIST 1.1-measureable disease or bone metastases only or bone-predominant disease received pembrolizumab 200 mg via IV infusion
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 1 and 2 Combined | Cohorts 1, 2, and 3 Combined | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 133 | 67 | 58 | 81 | 45 | 200 | 258 | 126
Percentage of Participants | 10.5 [5.9 to 17.0] | 4.5 [0.9 to 12.5] | 24.1 [13.9 to 37.2] | 29.6 [20.0 to 40.8] | 31.1 [18.2 to 46.6] | 8.5 [5.0 to 13.3] | 12.0 [8.3 to 16.6] | 30.2 [22.3 to 39.0]

5. Secondary Outcome: Duration of Response (DOR) Per PCWG3-modified RECIST 1.1 (Cohort 1, Cohort 2, Cohort 4 and Cohorts 1 and 2 Combined)
Description: DOR was defined as the time from first documented evidence of complete response (CR; disappearance of all target lesions) or partial response (PR; ≥30% decrease in the sum of diameters of target lesions) until progressive disease (PD) assessed by central imaging where PD was determined by radionuclide bone scan using Prostate Cancer Working Group (PCWG3)-modified RECIST 1.1 criteria and PD for all other tumors was determined using RECIST 1.1 or death due to any cause, whichever occurred first. Per protocol, analysis for this outcome measure was conducted in Cohorts 1, 2 and 4 separately, well as in Cohorts 1 and 2 combined for the first course of treatment.
Time Frame: Up to ~52 months
Population: The analysis was based on all responders with measurable disease at baseline in the ASaT population which consisted of all allocated participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohorts 1 and 2 Combined
Number analyzed (Participants) | 8 | 2 | 10 | 10
Months | NA [1.9 to NA] — NA = median and upper limit not reached due to an insufficient number of responding participants with relapse | NA [4.4 to NA] — NA = median and upper limit not reached due to an insufficient number of responding participants with relapse | NA [NA to NA] — NA = median and lower and upper limits not reached due to an insufficient number of responding participants with relapse | NA [1.9 to NA] — NA = median and upper limit not reached due to an insufficient number of responding participants with relapse

6. Secondary Outcome: DOR- Per RECIST 1.1 (Cohort 1, Cohort 2, Cohort 4 and Cohorts 1 and 2 Combined)
Description: DOR was defined as the time from first documented evidence of complete response (CR; disappearance of all target lesions) or partial response (PR; ≥30% decrease in the sum of diameters of target lesions) ) until progressive disease (PD) assessed by central imaging where PD was determined by radionuclide bone scan using RECIST 1.1 and PD for all other tumors was determined using RECIST 1.1 or death due to any cause, whichever occurred first. Per protocol, analysis for this outcome measure was conducted in Cohorts 1, 2 and 4 separately, well as in Cohorts 1 and 2 combined for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohorts 1 and 2 Combined
Number analyzed (Participants) | 8 | 2 | 10 | 10
Months | NA [1.9 to NA] — NA = median and upper limit not reached due to an insufficient number of responding participants with relapse | NA [4.4 to NA] — NA = median and upper limit not reached due to an insufficient number of responding participants with relapse | NA [NA to NA] — NA = median and lower and upper limits not reached due to an insufficient number of responding participants with relapse | NA [1.9 to NA] — NA = median and upper limit not reached due to an insufficient number of responding participants with relapse

7. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate (By Each Cohort, Cohorts 1 and 2 Combined, Cohorts 1, 2, and 3 Combined and Cohorts 4 and 5 Combined)
Description: Percentage of participants who had PSA response defined as at least 50% decline from baseline measured twice at least 3 weeks apart. Per protocol, analysis for this outcome measure was conducted in Cohorts 1 and 2 combined, Cohorts 1, 2, and 3 combined, Cohorts 4 and 5 combined well as in Cohorts 1 to 5 for the first course of treatment.
Time Frame: Up to ~52 months
Population: Analysis population was the ASaT which consisted of all allocated participants who received at least one dose of study treatment and had a PSA measurement at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 1 and 2 Combined | Cohorts 1, 2, and 3 Combined | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 124 | 61 | 58 | 80 | 45 | 185 | 243 | 125
Percentage of Participants | 6.5 [2.8 to 12.3] | 8.2 [2.7 to 18.1] | 1.7 [0.0 to 9.2] | 16.3 [8.9 to 26.2] | 8.9 [2.5 to 21.2] | 7.0 [3.8 to 11.7] | 5.8 [3.2 to 9.5] | 13.6 [8.1 to 20.9]

8. Secondary Outcome: Time to PSA Progression (By Each Cohort, Cohorts 1 and 2 Combined, Cohorts 1, 2, and 3 Combined and Cohorts 4 and 5 Combined)
Description: Time to PSA progression was defined as the time from first day of study treatment to the date of PSA progression. Participants without PSA progression were censored at the last PSA assessment date. PSA progression was defined as the date that an increase of 25% or more and an absolute increase of 2 ng/mL or more from the nadir were documented. For participants who had a decline in PSA during treatment, PSA progression must have been confirmed by a second value 3 or more weeks later increased with respect to the nadir PSA. Per protocol, analysis for this outcome measure was conducted in Cohorts 1 and 2 combined, Cohorts 1,2, and 3 combined, Cohorts 4 and 5 combined well as in Cohorts 1 to 5 separately for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 1 and 2 Combined | Cohorts 1, 2, and 3 Combined | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 133 | 67 | 58 | 81 | 45 | 200 | 258 | 126
Months | 5.1 [4.2 to NA] — NA = upper limit not reached due to insufficient number of participants with an event | 6.2 [4.2 to 6.9] | 4.2 [4.2 to 4.6] | 5.6 [4.2 to 10.4] | 4.2 [4.2 to 6.2] | 6.2 [4.2 to 6.9] | 4.4 [4.2 to 6.2] | 4.4 [4.2 to 6.2]

9. Secondary Outcome: Radiographic Progression-free Survival (rPFS) - Per PCWG3-modified RECIST 1.1 (By Each Cohort, Cohorts 1 and 2 Combined, Cohorts 1, 2, and 3 Combined, and Cohorts 4 and 5 Combined)
Description: rPFS was defined as the time from first day of study treatment to the documented disease progression by central imaging vendor where PD in bone-only tumors was determined by radionuclide bone scan using PCWG3 criteria and PD for all other tumors were determined using RECIST 1.1 or death due to any cause, whichever occurs first. Per protocol, analysis for this outcome measure was conducted in Cohorts 1 and 2 combined, Cohorts 1,2, and 3 combined, Cohorts 4 and 5 combined well as in Cohorts 1 to 5 separately for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 5: Bone Metastases Only or Bone-predominant Disease: Participants with bone metastases only or bone predominant disease received pembrolizumab 200 mg via IV infusion
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 1 and 2 Combined | Cohorts 1, 2, and 3 Combined | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 133 | 67 | 58 | 81 | 45 | 200 | 258 | 126
Months | 2.1 [2.0 to 2.1] | 2.1 [2.0 to 3.2] | 3.7 [2.1 to 4.2] | 4.2 [2.5 to 6.0] | 4.4 [3.2 to 6.2] | 2.1 [2.0 to 2.1] | 2.1 [2.1 to 2.2] | 4.2 [3.7 to 6.0]

10. Secondary Outcome: Overall Survival (OS) (By Each Cohort, Cohorts 1 and 2 Combined, Cohorts 1, 2, and 3 Combined, Cohorts 4 and 5 Combined)
Description: OS was defined as the time from first day of study treatment to the time of death. Participants without documented death were censored at the date of the last follow up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. Per protocol, analysis for this outcome measure was conducted in Cohorts 1 and 2 combined, Cohorts 1,2, and 3 combined, Cohorts 4 and 5 combined well as in Cohorts 1 to 5 separately for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: PD-L1 Positive With Measurable Disease | Cohort 2: PD-L1 Negative With Measurable Disease | Cohort 3: Bone Metastases With Non-measurable Disease | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 1 and 2 Combined | Cohorts 1, 2, and 3 Combined | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 133 | 67 | 58 | 81 | 45 | 200 | 258 | 126
Months | 9.5 [6.4 to 11.9] | 7.9 [5.9 to 10.2] | 14.1 [10.8 to 17.6] | 17.6 [14.0 to 22.6] | 20.8 [14.1 to 28.9] | 8.1 [6.6 to 10.7] | 9.6 [7.9 to 12.4] | 18.9 [16.2 to 23.6]

11. Secondary Outcome: Duration of PSA Response (Cohorts 4 and 5 by Cohort and Combined)
Description: Duration of PSA response was defined as the time from PSA response, when the PSA value first declined by at least 50% of the baseline (must have been confirmed by a second value), to the date of PSA progression at which there was an increase of 25% or more from the nadir PSA, provided the absolute increase from the nadir PSA was at least 2 ng/mL. Per protocol, analysis for this outcome measure was conducted in Cohorts 4 and 5 separately and combined for the first course of treatment.
Time Frame: Up to ~52 months
Population: Analysis population was the ASaT which consisted of all allocated participants who received at least 1 dose of study treatment and had a confirmed PSA response.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 13 | 4 | 17
Months | 8.3 [2.8 to NA] — NA = Upper limit was not reached due to no progressive disease by the time of last disease assessment | 18.0 [3.0 to NA] — NA = Upper limit was not reached due to no progressive disease by the time of last disease assessment | 18.0 [2.8 to NA] — NA = Upper limit was not reached due to no progressive disease by the time of last disease assessment

12. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy (Cohorts 4 and 5 by Cohort and Combined)
Description: Time to initiation of cytotoxic chemotherapy was defined as the time from first day of study treatment to the time of initiation of cytotoxic chemotherapy for prostate cancer. The median time was calculated using the Kaplan-Meier method for censored data. Per protocol, analysis for this outcome measure was conducted in Cohorts 4 and 5 separately and combined for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 81 | 45 | 126
Months | 11.1 [8.5 to 17.4] | 11.3 [9.0 to 14.5] | 11.1 [9.4 to 14.5]

13. Secondary Outcome: Time to New-Anticancer Therapy (Cohorts 4 and 5 By Cohort and Combined)
Description: Time to new-anticancer therapy was defined as the time from first day of study treatment to the time of new-anticancer therapy for prostate cancer. The median time was calculated using the Kaplan-Meier method for censored data. Per protocol, analysis for this outcome measure was conducted in Cohorts 4 and 5 separately and combined for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 81 | 45 | 126
Months | 9.5 [7.2 to 11.1] | 9.5 [5.9 to 11.5] | 9.5 [7.8 to 11.1]

14. Secondary Outcome: Time to First Skeletal-related Event (Cohorts 4 and 5 By Cohort and Combined)
Description: Time to initiation of first skeletal-related event was defined as the time from first day of study treatment to the first skeletal-related event, which was defined as radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression, or change or antineoplastic therapy to treat bone pain. Per protocol, analysis for this outcome measure was conducted in Cohorts 4 and 5 separately and combined for the first course of treatment.
Time Frame: Up to ~52 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 4: RECIST 1.1-measureable Disease | Cohort 5: Bone Metastases Only or Bone-predominant Disease | Cohorts 4 and 5 Combined
Number analyzed (Participants) | 81 | 45 | 126
Months | NA [27.6 to NA] — NA = median and upper limit of the 95% CI were not reached due to insufficient number of participants with an event | NA [NA to NA] — NA = median, lower and upper limits of the 95% CI were not reached due to insufficient number of participants with an event | NA [NA to NA] — NA = median, lower and upper limits of the 95% CI was not reached due to insufficient number of participants with an event

ADVERSE EVENTS:
Time Frame: Up to ~52 months
Description: All-Cause Mortality included all allocated participants. Serious and Other AEs were reported according to treatment course for all participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug were excluded as AEs.
Groups:
- Cohort 1 - First Course: Participants with PD-L1-positive, measurable disease received pembrolizumab 200 mg via IV infusion
- Cohort 2- 1st Course: Participants with PD-L1 negative, measurable disease received pembrolizumab 200 mg via IV infusion
- Cohort 3 - First Course: Participants with bone metastases and non-measurable disease received pembrolizumab 200 mg via IV infusion
- Cohort 4 - First Course: Participants with RECIST 1.1-measureable disease received pembrolizumab 200 mg via IV infusion
- Cohort 5 - First Course: Participants with bone metastases only or bone-predominant disease received pembrolizumab 200 mg via IV infusion
- Cohort 1 - Second Course: Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
Arm/Group | Cohort 1 - First Course | Cohort 2- 1st Course | Cohort 3 - First Course | Cohort 4 - First Course | Cohort 5 - First Course | Cohort 1 - Second Course
All-Cause Mortality (participants affected / at risk) | 126/133 | 63/69 | 57/58 | 76/81 | 40/47 | 0/1
Serious Adverse Events (participants affected / at risk) | 70/133 | 28/67 | 25/58 | 26/81 | 19/45 | 0/1
Other Adverse Events (participants affected / at risk) | 128/133 | 62/67 | 57/58 | 79/81 | 42/45 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - First Course (N=133) | Cohort 2- 1st Course (N=67) | Cohort 3 - First Course (N=58) | Cohort 4 - First Course (N=81) | Cohort 5 - First Course (N=45) | Cohort 1 - Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 3 (3) | 3 (3) | 2 (3) | 3 (4) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24) | 8 (8) | 7 (7) | 5 (5) | 4 (4) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Miller Fisher syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subdural hygroma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 10 (10) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perinephric collection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - First Course (N=133) | Cohort 2- 1st Course (N=67) | Cohort 3 - First Course (N=58) | Cohort 4 - First Course (N=81) | Cohort 5 - First Course (N=45) | Cohort 1 - Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 35 (39) | 12 (12) | 21 (24) | 11 (13) | 6 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (5) | 1 (1) | 1 (1) | 12 (12) | 8 (8) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 14 (15) | 7 (7) | 1 (1) | 6 (6) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 25 (27) | 21 (23) | 13 (15) | 12 (13) | 8 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 28 (35) | 17 (25) | 10 (12) | 24 (27) | 11 (15) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 6 (6) | 1 (1) | 9 (9) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 37 (45) | 26 (31) | 13 (15) | 19 (21) | 8 (9) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (22) | 18 (24) | 4 (4) | 5 (5) | 4 (4) | 1 (1)
Asthenia (General disorders) | 18 (20) | 11 (11) | 12 (14) | 9 (9) | 5 (5) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Chills (General disorders) | 7 (7) | 5 (5) | 1 (4) | 3 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 39 (41) | 22 (22) | 18 (18) | 36 (42) | 18 (19) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 4 (5) | 2 (2) | 4 (4) | 2 (2) | 7 (7) | 0 (0)
Malaise (General disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 21 (24) | 7 (8) | 5 (6) | 8 (12) | 3 (4) | 0 (0)
Pain (General disorders) | 4 (4) | 2 (2) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 13 (14) | 11 (13) | 3 (4) | 5 (5) | 3 (3) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 1 (1) | 3 (3) | 5 (7) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (14) | 5 (6) | 7 (8) | 6 (7) | 3 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 1 (1) | 12 (15) | 5 (10) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 1 (1) | 6 (6) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 11 (11) | 6 (6) | 6 (7) | 1 (1) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 4 (4) | 3 (5) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 8 (8) | 5 (5) | 4 (4) | 2 (3) | 4 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 6 (11) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 4 (6) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 16 (17) | 6 (6) | 9 (9) | 14 (15) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 38 (44) | 23 (25) | 19 (22) | 19 (23) | 11 (13) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 2 (2) | 7 (12) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 4 (8) | 2 (2) | 3 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9) | 4 (4) | 2 (2) | 7 (8) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (10) | 1 (1) | 4 (4) | 2 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (30) | 11 (11) | 9 (11) | 17 (23) | 8 (10) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (23) | 11 (12) | 13 (15) | 19 (20) | 15 (19) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (5) | 6 (6) | 0 (0) | 4 (5) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | 3 (3) | 7 (9) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4) | 7 (7) | 3 (4) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (13) | 7 (7) | 6 (6) | 12 (15) | 7 (8) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3) | 3 (3) | 8 (14) | 5 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3) | 4 (4) | 6 (7) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 5 (7) | 5 (6) | 5 (6) | 6 (6) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (9) | 4 (4) | 5 (6) | 5 (5) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 10 (18) | 3 (3) | 3 (3) | 9 (11) | 6 (7) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 5 (6) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 10 (11) | 4 (4) | 14 (14) | 5 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 6 (6) | 4 (4) | 11 (11) | 11 (12) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 0 (0) | 7 (7) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (16) | 4 (4) | 7 (7) | 16 (16) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 1 (1) | 19 (25) | 6 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 1 (1) | 9 (10) | 4 (5) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 6 (7) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 6 (9) | 0 (0) | 3 (4) | 9 (9) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have had the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must have been deleted prior to submission; this confidentiality did not include efficacy and safety results. Sponsor review could be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02787005/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT02787005/SAP_001.pdf